CLINICAL TRIAL: NCT05070052
Title: Comparing Mindfulness Based Cognitive Therapy to Cognitive Behavioral Therapy for Youth at High Risk for Mood and Psychotic Disorders: a Randomized Controlled Trial
Brief Title: MBCT and CBT for Youth at High Risk for Mood and Psychotic Disorders: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, David J. Miklowitz, Ph.D., Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-000391
Record Dates: First submitted 2021-07-20; First posted 2021-10-06 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Mood Disorders; Prodromal Symptoms; Bipolar Disorder; Parents; Clinical High Risk
Keywords: group therapy; psychotherapy; psychoeducation; skills training; mood disorders; prodromal psychosis; adolescents; parent group; youth
MeSH Terms: conditions — Mood Disorders; Prodromal Symptoms; Bipolar Disorder | interventions — Cognitive Behavioral Therapy; Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group CBT (Experimental): 9 group sessions lasting 75-90 minutes each. CBT starts with psychoeducation about emotions, their primary functions, and how our emotions can affect the way we think and behave. They next learn about behavioral strategies that can help them manage or overcome difficult emotions. Group members also complete gradual exposure exercises, which involve engaging with activities that elicit negative emotions. Finally, group members are taught cognitive skills to help them cope with difficult/stressful thoughts.
  Interventions: Behavioral: cognitive behavioral therapy
- Group MBCT (Experimental): 9 group sessions lasting 75-90 minutes each. The focus of sessions 1 through 4 will be learning to bring greater awareness to the present moment, on purpose, and nonjudgmentally. Appropriate responding is the focus of sessions 5 through 8. All skills are reviewed in session 9.
  Interventions: Behavioral: mindfulness-based cognitive therapy

INTERVENTIONS:
Behavioral: cognitive behavioral therapy — 9 sessions of CBT weekly treatment in group setting
  Arms: Group CBT
Behavioral: mindfulness-based cognitive therapy — 9 sessions of MBCT weekly treatment in group setting
  Arms: Group MBCT

SUMMARY:
The present study is a randomized controlled trial comparing the efficacy and acceptability of CBT and MBCT group-based interventions adapted for young people at elevated risk for mood or psychotic disorder onset or relapse. Young people (ages 13-24) are provided with targeted psychoeducation and learn a variety of coping skills and wellness practices for mood regulation and stress and distress management. Parents meet separately to learn the same skills and receive guidance in supporting their youth with skill development. The therapy is also augmented by a mobile phone application that supports regular symptom monitoring and skills practice.

DETAILED DESCRIPTION:
Psychosocial interventions that improve emotional health and stability could have a dramatically favorable impact on individual suffering among adolescents and young adults at risk for severe mental illness, as well as their family members. Unfortunately, youth who are at risk for bipolar disorder or psychosis are treated with a wide variety of medications and therapies, with little evidence-based practice.

The main objective of this study is to investigate the comparative efficacy and acceptability of weekly outpatient group-based Mindfulness based Cognitive Therapy (MBCT) and Cognitive Behavioral Therapy (CBT) adapted for youth at elevated risk for serious or persistent mood disorders or psychosis. Consistent with the National Institute of Mental Health's shift towards common underlying mechanisms across diagnoses ("Research Domain Criteria, or RDoc; Sanislow et al., 2010), recruitment for this study is transdiagnostic, targeting a range of youth with difficulties with mood dysregulation and stress.

All randomized control trial (RCT) participants receive one of the two active treatments. The order of treatment groups has been randomized, with participants blinded to their treatment assignment. Five to 15 young participants of similar age (teen or young adult) comprise each group. Parents receive a parallel parent-only group that informs them of the content and skills presented to their offspring.

The investigators will assess emotion dysregulation, psychiatric symptoms, overall functioning, and quality of life at baseline, immediately following the 9-week treatment, and at follow-up (3 months after therapy ends).

Clinical symptoms, cognitions, mindfulness, emotion regulation, and well-being will be measured at baseline and each follow-up assessment. Both youth and young adults will participate in a follow-up assessment immediately after the intervention. Youth participants will participate in a second follow-up assessment 12 weeks post-treatment.

The main investigative hypotheses are that both the MBCT and CBT programs will be acceptable to the young participants and parents and associated with high satisfaction ratings. Additionally, the investigators anticipate that both MBCT and CBT will be associated with comparable improvements in mood, anxiety, and psychotic symptoms and social functioning from pretreatment to final follow-up. Finally, the investigators anticipate that increases in mindfulness and reductions in negative cognitions from pretreatment to post-treatment and follow-up will be correlated with improvements in the young participants' self-reported emotional dysregulation and attention.

The study aims to add to the body of knowledge on evidence-based interventions targeting mood and stress pathways for youth at risk for chronic or serious mental health challenges.

ELIGIBILITY:
Inclusion Criteria:

- Patient meets criteria for having experienced a (past or present) disorder marked by clinically significant mood instability, depression, and/or psychotic features (i.e., diagnosed with a mood disorder, adjustment disorder with depressed mood, or psychotic disorder) OR they are at clinical high risk for psychosis

Exclusion Criteria:

* Patient's current severity of illness interferes with participation in a group treatment (e.g., preoccupied with internal stimuli)
* Patient has a current substance use disorder
* Patient has a pervasive developmental disorder or intellectual disability
* Patient cannot speak and read English sufficiently to allow for valid interpretation of a clinical assessment provided in English

Ages: 9 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Children's Depression Rating Scale-Revised (CDRS-R; Poznanski & Mokros, 1996) scores at 9 weeks & 6 months. | 0 & 9 weeks, 6 months
  Semi-structured interview of youth and parent to assess recent severity of youth depression. Consensus scores are obtained for 17 items, with total scores ranging from 17 to 113 and higher scores indicating more severe depression.
Change from Baseline in Questionnaire for Measuring Health-Related Quality of Life in Children (KINDL; Ravens-Sieberer & Bullinger, 1998) scores at 9 weeks & 6 months | 0 & 9 weeks, 6 months
  Self-report measure of health-related quality of life in children and adolescents. Both the parent-report scale (24-item) & adolescent-report scale (31-item) are included, with higher total scale scores (range 0 to 100) indicating more severe problems with health-related quality of life.
Change from Baseline Children's Global Assessment Scale (C-GAS; Shaffer, 1983) scores at 9 weeks & 6 months | 0 & 9 weeks, 6 months
  Assessor-rated rating of current global functioning, considering illness severity. Scores range from 1 to 100, with higher scores indicating better global functioning.
Change from Baseline Young Mania Rating Scale (YMRS; Young, Biggs, Ziegler, & Meyer, 1978) scores at 9 weeks & 6 months | 0 & 9 weeks, 6 months
  Semi-structured interview of youth and parent on recent manic mood symptoms. Consensus scores are obtained from 11 items, with total scale scores ranging from 0 to 60 and higher scores indicating more severe manic symptoms.
Change from Baseline Prodromal Questionnaire - Brief (PQ-B; Loewy, Pearson, Vinogradov, Bearden, & Cannon, 2011) scores at 9 weeks & 6 months | 0 & 9 weeks, 6 months
  Patient self-report measure of current severity of positive clinical high risk for psychosis symptoms. Total score is based on 21 items and represents higher level of positive symptomatology, considering associated distress and impact.

SECONDARY OUTCOMES:
Change from Baseline Difficulties in Emotion Regulation Scale (DERS; Gratz & Roemer, 2004) scores at 9 weeks & 6 months | 0 & 9 weeks, 6 months
  Parental self-report measure of their own difficulties in emotion regulation. Total scores on this 36-item instrument range from 36 to 180, with higher scores indicating more severe personal difficulties with emotion regulation.
Change from Baseline Depression Anxiety Stress Scales-21 (DASS-21; Lovibond & Lovibond, 1995) scores at 9 weeks & 6 months | 0 & 9 weeks, 6 months
  Parental self-report measure of their own difficulties with depression, anxiety and stress. Total scores on this 21-item instrument range from 0 to 63, with higher scores indicating more severe personal difficulties with emotion regulation.
Change from Baseline Brief COPE Inventory (Brief-COPE; Carver, 1997) scores at 9 weeks & 6 months | 0 & 9 weeks, 6 months
  Youth self-report measure of their use of emotional behavioral coping strategies for stressful situations. Scores for the 28-item measure range from 28 to 112, with higher scores indicating greater use of coping strategies.

CONTACTS AND LOCATIONS:
Overall Officials: David Miklowitz, PhD, Principal Investigator — University of California, Los Angeles; Danielle M. Denenny, PhD, Study Director — University of California, Los Angeles; Marc J. Weintraub, Study Director — University of California, San Diego
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weintraub MJ, Denenny D, Ichinose MC, Zinberg J, Morgan-Fleming G, Done M, Brown RD, Bearden CE, Miklowitz DJ. A randomized trial of telehealth mindfulness-based cognitive therapy and cognitive behavioral therapy groups for adolescents with mood or attenuated psychosis symptoms. J Consult Clin Psychol. 2023 Apr;91(4):234-241. doi: 10.1037/ccp0000782. Epub 2023 Jan 16. PMID 36649157